CLINICAL TRIAL: NCT02154919
Title: Conservative Pharmacotherapy Versus Staged Percutaneous Coronary Intervention on Non-culprit Vessels for ST-Segment Elevation Myocardial Infarction Patients With Multivessel Disease
Brief Title: Non-culprit Vessels for ST-Segment Elevation Myocardial Infarction
Acronym: CPVsSPCI
Status: Completed | Type: Observational
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Peng Jian Jun, Beijing Shijitan Hospital, Capital Medical University , Beijing, China, Beijing Shijitan Hospital, Capital Medical University
Other Study IDs: CPVsSPCI
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Conservative Pharmacotherapy; Staged Percutaneous Coronary Intervention; Non-culprit Vessels; ST-Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- complete revascularization group: this group underwent second PCI procedure on the non-culprit vessels and reveived 100-120 IU/kg unfractionated heparin during PPCI, followed by 3 days administration of low molecular weight heparin or Fondaparinux sodium after procedure. Patients in the CP group and CR group after second PCI procedure were given conservative medicine such as Statins which were not contraindicated to the patients.
  Interventions: Procedure: Percutaneous coronary intervention
- conservative pharmacotherapy group: patients in conservative group undergoing pharmacotherapy after PPCI. The drugs were the same between two groups.

INTERVENTIONS:
Procedure: Percutaneous coronary intervention
  Groups: complete revascularization group

SUMMARY:
To compare the different effect of conservative pharmacotherapy and Staged Percutaneous Coronary Intervention (SPCI) on significant non-culprit lesions in patients with ST-segment elevation myocardial infarction (STEMI) at presentation remains controversial

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 75 with continuous ischemic chest pain for ≥ 30 minutes and ST-segment of electrocardiographic leads between V2 and V3 elevated ≥ 0.2 mV (or ≥ 0.1 mV in ≥ 2 other continuous electrocardiographic leads), cardiac troponin I (cTn I) elevation of > 0.05 ng/ml, coronary arteriography within 12 hours after the onset of symptoms indicating lesion in culprit vessel with thrombolysis in myocardial infarction (TIMI) flow grade 0 to 1, merely underwent PPCI. Additionally, coronary arteriography corroborates lesions in non-culprit vessel (Besides the culprit vessel, there are ≥ 70% stenoses in one or more coronary vessels in which diameters were ≥ 2 mm).

Exclusion Criteria:

* left main coronary artery disease, cardiogenic shock, complete left bundle branch block (CLBBB) PPCI treated culprit and non-culprit vessels, PPCI failure patients with postsurgical haemodynamic instability or spontaneous ischemia, ≥ 70% stenoses of vessels remained during the hospitalization after staged PCI, history of PCI or Coronary Artery Bypass Grafting (CABG), history of chronic cardiac failure, bleeding diathesis, prior administration of thrombolytic therapy, known thrombopenia or leucopenia, sever liver and kidney dysfunction, active infection, immune system and connective tissue diseases, known contraindications to aspirin or heparin, life expectancy < 1 year, had major procedure within 3 months, uncontrolled hypertension, ischemic stroke within 30 days, hemorrhagic stroke, intracranial diseases including and arteriovenous malformation, extensive traumatic cerebral infarction within 6 weeks, oral anticoagulant therapy, severe myocardial infarction related complications and perioperative death

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients after culprit vessels treated by PPCI
Sampling Method: Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 360days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China